CLINICAL TRIAL: NCT00788554
Title: LEVEL Trial: Correction of Inguinal Hernia, Endoscopic Versus Lichtenstein. A Randomised Controlled Clinical Trial.
Brief Title: LEVEL Trial: Correction of Inguinal Hernia, Endoscopic Versus Lichtenstein
Acronym: LEVEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, hasan eker, Prof. Dr. J.F. Lange, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEVEL
Record Dates: First submitted 2008-11-09; First posted 2008-11-11 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Inguinal Hernia
Keywords: groin; inguinal; hernia; lichtenstein; TEP
MeSH Terms: conditions — Hernia, Inguinal; Hernia | interventions — tetraethylpyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: Lichtenstein procedure
- 2 (Active Comparator)
  Interventions: Procedure: TEP

INTERVENTIONS:
Procedure: Lichtenstein procedure — open surgical procedure for inguinal hernia correction
  Arms: 1
Procedure: TEP — Total Exta Peritoneal procedure for inguinal hernia correction
  Arms: 2

SUMMARY:
The aim of this study is to compare laparoscopic total extraperitoneal and open mesh repair of inguinal hernia, with regard to hospital stay, postoperative pain, quality of life, postoperative recovery and return to daily activities, complications and recurrences

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age > 18 years
* inguinal hernia(primary, recurrence or bilateral)
* elective procedure

Exclusion Criteria:

* Scrotal hernia
* Prostatectomy, Pfannenstiehl-incision, pre-peritoneal surgery in history
* Participation in other trial
* Pregnancy
* Communicative or cognitive restrictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2000-08; Primary Completion 2004-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
hospital stay | 7 days
postoperative pain | 6 weeks
return to work | 6 weeks
quality of life | 5 years

SECONDARY OUTCOMES:
operating time | 1 day
operating costs | 1 week
complication | 1 month
mortality | 5 years
total costs | 1 month
recurrence | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: J.F. Lange, professor, Principal Investigator — Erasmus Medical Center; J.J. Jeekel, professor, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Eker HH, Langeveld HR, Klitsie PJ, van't Riet M, Stassen LP, Weidema WF, Steyerberg EW, Lange JF, Bonjer HJ, Jeekel J. Randomized clinical trial of total extraperitoneal inguinal hernioplasty vs Lichtenstein repair: a long-term follow-up study. Arch Surg. 2012 Mar;147(3):256-60. doi: 10.1001/archsurg.2011.2023. PMID 22430907
- [Derived] Langeveld HR, van't Riet M, Weidema WF, Stassen LP, Steyerberg EW, Lange J, Bonjer HJ, Jeekel J. Total extraperitoneal inguinal hernia repair compared with Lichtenstein (the LEVEL-Trial): a randomized controlled trial. Ann Surg. 2010 May;251(5):819-24. doi: 10.1097/SLA.0b013e3181d96c32. PMID 20395851